CLINICAL TRIAL: NCT00053677
Title: Naltrexone Treatment in Pathologic Gambling Disorder
Brief Title: Drug Treatment for Pathologic Gambling Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21MH065920 (NIH); R21MH065920 (NIH); DSIR AT-AS
Record Dates: First submitted 2003-02-04; First posted 2003-02-05 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Gambling
Keywords: Impulse Control Disorders
MeSH Terms: conditions — Gambling; Disruptive, Impulse Control, and Conduct Disorders | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Naltrexone (Placebo Comparator): 17 weeks of double-blind Naltrexone. Subjects were randomized into one of these three conditions (if they weren't randomized to placebo): naltrexone 50mg/day, 100mg/day, 150mg/day. To minimize nausea, treatment for all subjects was initiated at 25mg/day naltrexone for two days, then the dose was increased to 50mg/day. At week 3, subjects were randomly assigned to 50mg/day continued at that dose, while subjects who were randomized to naltrexone 100mg/day or 150mg/day were raised to the higher doses.
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Subjects who were assigned to placebo in the 17 week double-blind phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — For subjects who were randomly assigned to naltrexone 50mg/day, 100mg/day, or 150mg/day.
  Arms: Naltrexone
Drug: Placebo — For subjects who were randomly assigned to placebo.
  Arms: Placebo

SUMMARY:
This study will establish the best dose of the drug naltrexone to treat patients with Pathological Gambling Disorder (PGD) and severe urge symptoms.

DETAILED DESCRIPTION:
PGD is a prominent and growing social problem. Unfortunately, there is no established drug treatment for this disorder. Preliminary investigations demonstrate that naltrexone in doses up to 250 mg/day is well tolerated and safe during an 11-week period and may be a viable treatment option for PGD patients with severe urges. The implications of this study extend from PGD to other impulse control disorders, including compulsive shopping, kleptomania, and possibly alcoholism.

Participants are randomly assigned to receive either naltrexone or placebo for 16 weeks. The responses of men and women are compared to determine whether efficacy is distributed in a male:female ratio analogous to that of the PGD population in the United States. A Clinical Global Impression and a Gambling Symptom Scale are used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual IV criteria for Pathological Gambling Disorder
* Moderate or severe gambling urge assessed by the Gambling Symptom Assessment Scale
* No psychiatric drug use for 2 weeks or more
* Score >= 5 on The South Oaks Gambling Screen
* Hamilton Depression Rating Scale and Anxiety Rating score < 26. An increase (up to 10 points) of the scores is allowed unless the subject shows the risks of suicide.
* Completion of complete blood count, urinalysis, liver and thyroid function tests, and pregnancy tests, with no evidence of significant lab abnormalities
* Reliable birth control in women of child-bearing potential

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2002-12; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suck Won Kim, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical School, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Kim SW, Grant JE, Adson DE, Shin YC. Double-blind naltrexone and placebo comparison study in the treatment of pathological gambling. Biol Psychiatry. 2001 Jun 1;49(11):914-21. doi: 10.1016/s0006-3223(01)01079-4. PMID 11377409
- [Background] Kim SW. Opioid antagonists in the treatment of impulse-control disorders. J Clin Psychiatry. 1998 Apr;59(4):159-64. PMID 9590665
- [Background] Kim SW, Grant JE. An open naltrexone treatment study in pathological gambling disorder. Int Clin Psychopharmacol. 2001 Sep;16(5):285-9. doi: 10.1097/00004850-200109000-00006. PMID 11552772
- [Background] Grant JE, Kim SW. Demographic and clinical features of 131 adult pathological gamblers. J Clin Psychiatry. 2001 Dec;62(12):957-62. doi: 10.4088/jcp.v62n1207. PMID 11780876
- [Background] Kim SW, Grant JE. Personality dimensions in pathological gambling disorder and obsessive-compulsive disorder. Psychiatry Res. 2001 Nov 30;104(3):205-12. doi: 10.1016/s0165-1781(01)00327-4. PMID 11728609
- [Background] Kim SW, Grant JE. The psychopharmacology of pathological gambling. Semin Clin Neuropsychiatry. 2001 Jul;6(3):184-94. doi: 10.1053/scnp.2001.22924. PMID 11447570
- See also: Related Info — http://www.impulsecontroldisorders.org/index.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 83 participants began the placebo lead-in phase. 6 of those were placebo responders. The remaining 77 were randomized to Naltrexone or placebo.
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 58 | 19
Completed | 36 | 13
Not Completed | 22 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 58 | 19 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.8 (9.65) | 44.7 (9.67) | 46.3 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 10 | 47
  Male | 21 | 9 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 54 | 16 | 70
  Race/Ethnicity: Other Race | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 58 | 19 | 77

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive Compulsive Scale for Pathological Gambling (PG-YBOCS)
Description: A gambling severity measure derived from the Yale-Brown Obsessive Compulsive Scale. It sums gambling urges and thoughts questions to make a total score. Total scores range from 0 to 40, which higher scores indicating more severe gambling symptoms (worse outcome).Administered every week for the first 8 weeks and every other week for the remaining 10 weeks. Final visit scores were the scores measured at the last visit for each participant; data from previous visits were not combined to compute this value.
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 58 | 19
units on a scale
  Baseline | 16.9 (6.60) | 18.6 (4.90)
  Final Visit Score | 9.7 (8.12) | 12.9 (9.31)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the study (18 weeks per subject).
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/19
Other Adverse Events (participants affected / at risk) | 50/58 | 17/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=58) | Placebo (N=19)
Headache (Nervous system disorders) | 23 | 9
Nausea (Gastrointestinal disorders) | 35 | 7
Diarrhea (Gastrointestinal disorders) | 8 | 6
Constipation (Gastrointestinal disorders) | 3 | 3
Dry Mouth (General disorders) | 8 | 2
Dizziness (General disorders) | 6 | 1
Insomnia (Nervous system disorders) | 7 | 0

LIMITATIONS AND CAVEATS:
Pathological gambling is a chronic disease that may require long-term therapy. Although this study is one of the longest medication trials for PG, the study did not assess treatment effects beyond the acute 18-week treatment period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No